CLINICAL TRIAL: NCT04868539
Title: Influence of Nocturnal Light Exposure on the Impairment of Glucose Tolerance Induced by Chronic Sleep Restriction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Charles A. Czeisler, PhD, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2021P000961
Record Dates: First submitted 2021-04-20; First posted 2021-05-03 (Actual); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Glucose Intolerance; Sleep Deprivation; Sleep
Keywords: Chronic Sleep Restriction; Artificial Light At Night; Glucose Intolerance; Melatonin; Sleep
MeSH Terms: conditions — Glucose Intolerance; Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: This study uses a within-subjects randomized crossover design to compare the effects of sleep restriction with and without ALAN on glucose metabolism. The order in which subjects undergo the two sleep interventions will be randomized.
Who Masked: Participant
Masking Description: The order in which subjects undergo the two sleep interventions will be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Restriction with ALAN, then Sleep Restriction without ALAN (Experimental): Participants first received Sleep Restriction with extended duration Artificial Light At Night (ALAN), during which sleep episodes were shortened to 5 hours and participants remained in room lighting for the full wake episode (19h room light, 5h darkness). After a washout of 10 days, participants received Sleep Restriction without ALAN, during which sleep episodes were shortened to 5 hours but participants were kept in dim light for the extra time awake (14h room light, 5h dim light, 5h darkness).
  Interventions: Other: Sleep Restriction with ALAN first, then Sleep Restriction without ALAN
- Sleep Restriction without ALAN, then Sleep Restriction with ALAN (Experimental): Participants first received Sleep Restriction without extended duration Artificial Light At Night (ALAN), during which sleep episodes were shortened to 5 hours but participants were kept in dim light for the extra time awake (14h room light, 5h dim light, 5h darkness). After a washout of 10 days, participants received Sleep Restriction with extended duration ALAN, during which sleep episodes were shortened to 5 hours and participants remained in room lighting for the full wake episode (19h room light, 5h darkness).
  Interventions: Other: Sleep Restriction without ALAN first, then sleep restriction with ALAN

INTERVENTIONS:
Other: Sleep Restriction with ALAN first, then Sleep Restriction without ALAN — Sleep restriction with 90 lux lighting for 19hr/day first, followed by Sleep restriction with 90 lux lighting for 14hr/day
  Other Names: ALAN first
  Arms: Sleep Restriction with ALAN, then Sleep Restriction without ALAN
Other: Sleep Restriction without ALAN first, then sleep restriction with ALAN — Sleep restriction with 90 lux lighting for 14hr/day first, followed by Sleep restriction with 90 lux lighting for 19hr/day
  Other Names: ALAN second
  Arms: Sleep Restriction without ALAN, then Sleep Restriction with ALAN

SUMMARY:
This project is designed to test for the first time whether glucose metabolism is differentially impaired by sleep restriction with and without additional exposure to artificial light at night (ALAN).

DETAILED DESCRIPTION:
Laboratory studies have shown that sleep restriction to 4-6h per night for durations varying from one to 14 days reduces glucose tolerance in otherwise healthy adults, but the mechanisms by which insufficient sleep impairs glucose metabolism are still unknown. Current theories are based on the premise that the adverse metabolic consequences are caused by reduction in the duration of sleep per se. However, sleep curtailment is typically accompanied by longer exposure to artificial light at night (ALAN), which is an environmental endocrine disrupter that profoundly disrupts circadian rhythms.

The investigators have previously reported that acute circadian misalignment induced hyperglycemia comparable to pre-diabetic states in a third of otherwise healthy participants. Since then, the investigators have shown that even when the circadian phase of participants was realigned, prior exposure to 2 ½ weeks of chronic sleep restriction combined with a history of recurrent circadian disruption induced even more deleterious effects on glucose metabolism, in which pancreatic beta cells failed to respond adequately to increased glucose levels. Moreover, both night and rotating shift work (which induce circadian disruption) are associated with increased risk for metabolic problems. Night shifts can lead to acute increases in glucose and insulin levels, although some studies report reduced insulin release in response to meals consumed during the night. Given that circadian disruption has been shown to independently adversely affect metabolism, and exposure to ALAN adversely impacts metabolism in animals, it is important to understand the extent to which circadian disruption contributes to the observed impact of sleep curtailment on metabolism. No previous studies of the metabolic impact of sleep restriction in humans have controlled for this additional exposure to ALAN, thus confounding the effects of sleep restriction with the effects of circadian disruption caused by extended exposure to ALAN.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults with conventional and regular sleep-wake timing
* Non-smokers
* Completion of medical, psychological, and sleep screening tests
* Able to spend 33 consecutive days/nights in the laboratory
* Normal color vision

Exclusion Criteria:

* History of neurological or psychiatric disorder
* History of sleep disorder or regular use of sleep-promoting medication
* Current prescription, herbal, or over-the-counter medication use
* Traveling across 2 or more time zones within past 3 months
* Donating blood within past 8 weeks
* Worked night or rotating shift work within past 3 years
* Hearing impairment, visual impairment
* History of eye trauma or surgery
* Drug or alcohol dependency

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles A Czeisler, PhD, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteers were recruited through online advertisements between October 2021-December 2023.
Pre-assignment Details: Two participants were excluded prior to randomization; one was due to an undisclosed surgery that excluded them from the study, and the other was due to ending study enrollment before they were admitted.
Period: Overall Study
Arm/Group | Sleep Restriction With ALAN, Then Sleep Restriction Without ALAN | Sleep Restriction Without ALAN, Then Sleep Restriction With ALAN
Started | 6 | 6
Completed | 5 | 5
Not Completed | 1 | 1
Not completed — Unable to complete study due to poor IV access | 1 | 1

BASELINE CHARACTERISTICS:
Population: 10 participants were included in analyses. We were unable to obtain baseline measures for 2 participants who were randomized but did not complete. We were also unable to perform the IVGTT in 1 participant in the Sleep Restriction without ALAN, then Sleep Restriction with ALAN group so analyzed only 4 participants for outcome measures which used minimal model analysis. For other outcomes (e.g. melatonin duration and glucose tolerance), all 5 participants in this group were included.
Groups:
- Sleep Restriction With ALAN, Then Sleep Restriction Without ALAN: Participants first received Sleep Restriction with extended duration Artificial Light At Night (ALAN), during which sleep episodes were shortened to 5 hours and participants remained in room lighting for the full wake episode (19h room light, 5h darkness). After a washout of 10 days, participants received Sleep Restriction without extended duration Artificial Light At Night (ALAN), during which sleep episodes were shortened to 5 hours but participants were kept in dim light for the extra time awake (14h room light, 5h dim light, 5h darkness).
- Total: Total of all reporting groups
Arm/Group | Sleep Restriction Without ALAN, Then Sleep Restriction With ALAN | Sleep Restriction With ALAN, Then Sleep Restriction Without ALAN | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 3 | 3 | 6
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Impairment of Insulin Sensitivity
Description: Insulin sensitivity (Si) is assessed via minimal model analysis, a mathematical model developed by Bergman and colleagues. Higher values represent better insulin sensitivity and lower values represent impaired insulin sensitivity.
  The mean change in Si between exposure and baseline is reported for each arm.
Time Frame: Change between Study Day 7 vs. Study Day 15 and Study Day 24 vs. Study Day 32
Population: One participant excluded from "Without ALAN" condition due to non-physiological assay results
Measure: Mean (Standard Deviation); unit: (mU/L)^-1 min^-1
Groups:
- ALAN: Participants exposed to sleep restriction with extended duration artificial light at night (ALAN) during study days 8-14 or 25-31
- Without ALAN: Participants exposed to sleep restriction without extended duration artificial light at night (ALAN) during study days 8-14 or 25-31
Arm/Group | ALAN | Without ALAN
Number analyzed (Participants) | 9 | 8
(mU/L)^-1 min^-1 | -0.80 (1.63) | 0.55 (4.18)

2. Primary Outcome: Impairment of Glucose Tolerance
Description: Test the hypothesis that exposure to one week of sleep restriction with concurrent exposure to extended duration ALAN (LD 19:5) will induce greater impairment of glucose tolerance than exposure to one week of sleep restriction without extended duration ALAN (LD 14:10). Glucose tolerance will be calculated as the area under the curve from minutes 0-120 following a mixed meal tolerance test
Time Frame: Change between Study Day 6 vs. Study Day 14 and Study Day 23 vs. Study Day 31
Measure: Mean (Standard Deviation); unit: mg/dL*min
Arm/Group | ALAN | Without ALAN
Number analyzed (Participants) | 8 | 8
mg/dL*min | 524.4 (376.7) | 179.1 (1121.6)

3. Primary Outcome: Duration of Nocturnal Melatonin Secretion
Description: Test the hypothesis that exposure to one week of sleep restriction with concurrent exposure to extended duration ALAN (LD 19:5) will acutely reduce the duration of nocturnal melatonin secretion as compared to baseline more than exposure to one week of sleep restriction without extended duration ALAN (LD 14:10). Duration of nocturnal melatonin secretion will be determined by the duration of time at which melatonin levels are above a threshold calculated as 25% of peak-to-trough amplitude at baseline in dim light.
Time Frame: Change between Study Day 14-15 (overnight) vs. Study Day 31-32 (overnight)
Population: Unable to calculate melatonin duration for one participant under the Without ALAN condition due to IV sampling difficulties
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | ALAN | Without ALAN
Number analyzed (Participants) | 10 | 9
minutes | 432.9 (90.3) | 579.6 (44.8)

4. Secondary Outcome: Acute Insulin Response to Glucose
Description: Acute Insulin Response as calculated with minimal model analysis, a mathematical model developed by Bergman and colleagues, and represents early insulin release in the body to manage blood glucose levels. Higher values represent a better response and lower values represent a worse response. The mean change in AIRg between exposure and baseline is reported for each arm.
Time Frame: Change from study day 7 to 15 compared to change from study day 24 to 32
Measure: Mean (Standard Deviation); unit: (mU/L)^-1 min^-1
Arm/Group | ALAN | Without ALAN
Number analyzed (Participants) | 9 | 9
(mU/L)^-1 min^-1 | -110.41 (472.51) | -37.04 (203.45)

5. Secondary Outcome: Glucose Effectiveness
Description: Glucose Effectiveness as calculated using minimal model analysis, a mathematical model developed by Bergman and colleagues. It represents how well the body can normalize blood glucose independent of insulin. Higher glucose effectiveness (Sg) is generally associated with better metabolic health outcomes.
Time Frame: Change from study day 7 to 15 vs change from study day 24 to 32
Measure: Mean (Standard Deviation); unit: min^-1
Arm/Group | ALAN | Without ALAN
Number analyzed (Participants) | 9 | 9
min^-1 | -0.00049 (0.0051) | -0.0012 (0.0073)

6. Secondary Outcome: Insulin Area-under-the-curve
Description: Insulin area under the curve (AUC) as calculated with trapezoidal method between 0-120min following mixed meal tolerance test.
Time Frame: Change between Study Day 6 vs. Study Day 14 and Study Day 23 vs. Study Day 31
Population: We were unable to obtain meal response data for 2 participants due to IV access issues.
Measure: Mean (Standard Deviation); unit: uIu/mL*min
Arm/Group | ALAN | Without ALAN
Number analyzed (Participants) | 8 | 8
uIu/mL*min | 663.4 (917.7) | -71.6 (702.5)

7. Secondary Outcome: Duration of Endogenous Melatonin Secretory Profile
Description: Test the hypothesis that exposure to one week of sleep restriction with concurrent exposure to extended duration ALAN (LD 19:5) will reduce the duration of the endogenous melatonin secretory profile more than exposure to one week of sleep restriction without extended duration ALAN (LD 14:10). Duration of nocturnal melatonin secretion will be determined by the duration of time at which melatonin levels are above a threshold calculated as 25% of peak-to-trough amplitude at baseline in dim light.
Time Frame: Study Day 15-16 vs Study Day 32-33
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | ALAN | Without ALAN
Number analyzed (Participants) | 10 | 10
minutes | 581.7 (51.1) | 609.6 (66.1)

ADVERSE EVENTS:
Time Frame: From admission to inpatient study until the participant's last inpatient day (up to 33 days)
Groups:
- Sleep Restriction With ALAN: Participants received Sleep Restriction with extended duration Artificial Light At Night (ALAN), during which sleep episodes were shortened to 5 hours and participants remained in room lighting for the full wake episode (19h room light, 5h darkness).
- Sleep Restriction Without ALAN: Participants received Sleep Restriction without extended duration Artificial Light At Night (ALAN), during which sleep episodes were shortened to 5 hours but participants were kept in dim light for the extra time awake (14h room light, 5h dim light, 5h darkness).
Arm/Group | Sleep Restriction With ALAN | Sleep Restriction Without ALAN
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 6/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Sleep Restriction With ALAN (N=12) | Sleep Restriction Without ALAN (N=12)
Headache (General disorders) | 1 (2) | 1/6 (5)
Lightheadedness (General disorders) | 0 | 2 (2)
Nausea (General disorders) | 0 | 1 (2)
Bruising/petechiae on arm (General disorders) | 0 | 1 (1)
Chest pressure (General disorders) | 1 (2) | 0
Stomach pain (General disorders) | 0 | 1 (2)

LIMITATIONS AND CAVEATS:
Study enrollment was ended early due to budgetary reasons, so we were unable to study the total number of participants planned. Thus, we may have limited statistical power to interpret the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-26): https://cdn.clinicaltrials.gov/large-docs/39/NCT04868539/Prot_SAP_000.pdf